CLINICAL TRIAL: NCT00948025
Title: A Multicenter, Prospective, Randomized, Comparative Study of Hollow Nerve Conduit and Avance Nerve Graft Evaluating Recovery Outcomes of Nerve Repair in the Hand. (CHANGE)
Brief Title: A Comparative Post-marketing Study of Commercially Available Peripheral Nerve Gap Repair Options
Acronym: CHANGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: transitioning from 361 HCT/P Tissue to a Biologic (BLA)
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANG-CP-004
Record Dates: First submitted 2009-07-17; First posted 2009-07-29 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Nerve Injury
Keywords: Peripheral Nerve Repair; Conduit; AVANCE; Neuroma Resection; Nerve Gap Repair; Digital Nerve Repair; Nerve Graft; Nerve Allograft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Avance Nerve Graft (Active Comparator): Commercially available Avance Nerve Graft for repair of nerve gap
  Interventions: Other: Processed Human Nerve Tissue
- Hollow Tube Conduit (Active Comparator): Commercially available hollow tube conduit for repair of nerve gap.
  Interventions: Device: Hollow tube nerve conduit, synthetic or biosynthetic

INTERVENTIONS:
Device: Hollow tube nerve conduit, synthetic or biosynthetic — Appropriately size matched hollow tube nerve conduit (Neurotube, NeuroLac, NeuraGen, NeuroMatrix, NeuroFlex)
  Other Names: Neurotube; NeuroLac; NeuraGen; NeuroMatrix; NeuroFlex
  Arms: Hollow Tube Conduit
Other: Processed Human Nerve Tissue — Implantation of appropriate length of processed human nerve tissue at time of surgery.
  Other Names: Avance Nerve Graft
  Arms: Avance Nerve Graft

SUMMARY:
This study is a comparison of sensory recovery outcomes following the use of AVANCE Nerve Graft or hollow tube conduit for peripheral nerve gap repairs in the hand.

DETAILED DESCRIPTION:
The CHANGE study is a post-marketing study designed as a prospective, single-blind, randomized, two phase study comparing clinical outcomes of AVANCE Nerve Graft to hollow tube conduits. The first phase (pilot phase) assesses projected differences expected between two treatment groups. The second phase of the study provides comparison data between the two treatment groups.

AVANCE Nerve Graft is current regulated in the United States as a 361 HCT/P Tissue for transplantation; not a Drug, Biologic, or Medical Device. Hollow tube conduits are currently regulated in the United States as medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Require primary or secondary nerve injury repair with Hollow Nerve Conduit or AVANCE™ in at least 1 digital nerve;
* Undergo End to End nerve to nerve graft coaptation on both the proximal and distal portion of the nerve gap in the AVANCE™ group or nerve entubulation in the Hollow Nerve Conduit group;
* Be willing to comply with all aspects of the treatment and evaluation schedule over a 12 Month duration; and
* Sign and date an IRB-approved written informed consent prior to initiation of any study procedures, including screening procedures.

Exclusion Criteria:

* Nerve gaps of < 5 mm or > 20 mm;
* Estimated distance of regeneration of >125 mm (distance from injury site to sensory target)
* Nerve crush or avulsion injuries;
* Incomplete nerve transections;
* Injury requiring replantation of target digit;
* Contralateral digital injuries corresponding to the target digit;
* Nerve injuries in the affected limb proximal to the crease of the wrist;
* End to side nerve repair;
* Injuries with significant vascular damage which may impair adequate perfusion of the target limb;
* Subjects who are undergoing treatment with chemotherapy, radiation therapy, or other know treatment which affects the growth of neural and/or vascular system;
* Use of bovine collagen based hollow nerve conduit in a subject with known or suspected bovine sensitivity;
* Subjects age ≤18 years or ≥70 years;
* History neuropathy, diabetic or any other known neuropathy;
* Secondary nerve repair >12 weeks post initial injury;
* Currently enrolled in another investigational study;
* Expected use of medications during the study that are known to cause peripheral neuropathy;
* History or Reynaud's or other disorder known to compromise circulation or sensation in the upper extremity; and
* Any subject who at the discretion of the Investigator is not suitable for inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erick W DeVinney, Study Director — Axogen Corporation
Locations (4):
- United States (4):
  - Georgia Hand, Shoulder and Elbow, Atlanta, Georgia
  - Indiana Hand Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Curtis National Hand Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
IPD will not be released to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 22 June 2009 and ended on 23 May 2012.
Groups:
- Avance Nerve Graft: Commercially available Avance Nerve Graft for repair of nerve gap
  Processed Human Nerve Tissue Scaffold: Implantation of appropriate length of processed human nerve tissue scaffold at time of surgery.
Period: Phase 1 (Pilot Phase)
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Started | 14 | 9
Completed | 5 | 6
Not Completed | 9 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Phase 2 (Comparative Phase)
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and received one of the study treatments (Safety Population).
Groups:
- Avance Nerve Graft: Commercially available Avance Nerve Graft for repair of nerve gap
  Processed Human Nerve Tissue: Implantation of appropriate length of processed human nerve tissue scaffold at time of surgery.
- Total: Total of all reporting groups
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 9 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 45 [21 to 63] | 39 [20 to 53] | 41 [20 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Recovery of Static 2-point Discrimination in the Affected Digit
Description: Mean change in static 2-Point Discrimination between baseline and 12 months
Time Frame: 12 Months
Population: Number of subjects
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 9
percent change from baseline | -65.6 (5.94) | -31.8 (10.90)
Statistical Analysis 1: Comparison: Avance Nerve Graft vs Hollow Tube Conduit; 1. P-value comparing static 2-point discrimination per visit derived from mixed linear modeling of longitudinal data. 2. P-Value is based on Mann-Whitney U test; Test type: Other — Mann-Whitney U test was used to derive p-values; p = 0.0433, Wilcoxon (Mann-Whitney) — 1. a priori threshold for statistical significance set at p<0.05. 2. the p-value was not adjusted for multiple comparisons

2. Secondary Outcome: Moving 2-point Discrimination
Description: Percent Change from Baseline of Moving 2-Point Discriminations at Month 12
Time Frame: 12 months
Population: Modified Intent-to-Treat Population (mITT): All participants who were randomized, received one of the study treatments, and completed at least the 3 month follow-up visit.
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 9
percentage
  Modified Intent to Treat population | -62.5 (4.78) | -35.4 (13.71)
  Per protocol population | -62.5 (4.78) | -35.4 (13.71)

3. Secondary Outcome: Semmes-Weinstein Monofilament Assessment
Description: Percent Change from Baseline of Semmes-Weinstein Monofilament Assessment at Month 12
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 9
percentage
  modified intent to treat | -46.1 (4.07) | -21.1 (6.66)
  per protocol | -46.1 (4.07) | -21.1 (6.66)

4. Secondary Outcome: 12-month DASH Core Module Scores
Description: Summary of Disability of the Arm, Shoulder, and Hand (DASH) scores (Core Module) at Month 12
  The Disabilities of the Arm, Shoulder and Hand (DASH) core module questionnaire is a 30-item questionnaire includes 21 physical function items, 6 symptom items, and 3 social/role function items. It is a patient reported questionnaire used to assess physical function and severity of symptoms in patients with musculoskeletal disorders of the upper limb. Each of the items in the DASH use a 5-point Likert scale to assess the corresponding severity or functional parameter. The outcome measure is scored based on the formula ([sum of n responses)/ - 30 (minimum score]/1.2 (range of scores ÷100), where n represents the number of completed items. Computed scores range from 0 (no disability) to 100 (most severe disability).
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 5 | 6
score on a scale
  modified intent to treat | 4.66 (2.90) | 7.77 (2.58)
  per protocol | 4.66 (2.90) | 7.77 (2.58)

5. Secondary Outcome: 12-month DASH (Work Module) Scores
Description: Summary of Disability of the Arm, Shoulder, and Hand (DASH) scores (Work Module) at Month 12
  The Disabilities of the Arm, Shoulder and Hand (DASH) Work Module questionnaire is a 4-item questionnaire used to identify the job-specific difficulties that workers might experience but which may not affect their activities of daily living. It is a patient reported questionnaire used to assess the impact that musculoskeletal disorders of the upper limb have on a patient's ability to perform work-related tasks. Each of the items in the DASH Work Module use a 5-point Likert scale to assess the corresponding severity or functional parameter. The outcome measure is scored based on the formula ([sum of n responses)/ - 4 (minimum score]/0.16 (range of scores ÷100), where n represents the number of completed items. Computed scores range from 0 (no difficulty) to 100 (most severe difficulty).
Time Frame: 12 month
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 4 | 6
score on a scale
  modified intent to treat | 0.00 (0.00) | 5.22 (4.09)
  per protocol | 0.00 (0.00) | 5.22 (4.09)

6. Secondary Outcome: 12- Month DASH (Sports/Performing Arts Module)
Description: Summary of Disability of the Arm, Shoulder, and Hand (DASH) scores (Sports/Performing Arts Module) at month 12
  The Disabilities of the Arm, Shoulder and Hand (DASH) Sports/Performing Arts Module questionnaire is a 4-item questionnaire used to identify the specific difficulties that professional athletes/performing artists might experience but which may not affect their activities of daily living. It is a patient reported questionnaire used to assess the impact that musculoskeletal disorders of the upper limb have on a patient's ability to perform sports or play a musical instrument. Each of the items in the DASH use a 5-point Likert scale to assess the corresponding severity or functional parameter. The outcome measure is scored based on the formula ([sum of n responses)/ - 4 (minimum score]/0.16 (range of scores ÷100), where n represents the number of completed items. Computed scores range from 0 (no difficulty) to 100 (most severe difficulty).
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 3 | 3
score on a scale
  modified intent-to-treat | 8.33 (8.33) | 18.77 (9.56)
  per protocol | 8.33 (8.33) | 18.77 (9.56)

7. Secondary Outcome: Pain at 12-months
Description: Summary of Pain Assessment using Visual Analogue Scale (VAS) at Month 12
  The Visual Analog Scale (VAS) For Pain is a patient reported outcomes scale whereby the patient indicates his/her current pain level by making a mark on a continuous horizontal 10 centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the subject is currently experiencing. VAS for Pain data are recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing no pain and 100 millimeters representing "the worst pain imaginable".
Time Frame: 12-months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 5 | 6
units on a scale
  modified intent to treat | 0.54 (0.28) | 0.92 (0.41)
  per protocol | 0.54 (0.28) | 0.92 (0.41)

8. Secondary Outcome: Thermal Discretion at 12-months
Description: Summary of Thermal Discretion at Month 12 as determined by the Investigator.
  Thermal discretion was assessed by applying a hot and/or cold object to the patient's affected digit. Thermal discretion was reported as either present ("Yes") or not present ("No").
Time Frame: 12-month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 7
Participants
  Modified Intent to Treat: Yes (Thermal Discretion) | 6 | 7
  Modified Intent to Treat: No (Thermal Discretion) | 0 | 0
  Per Protocol: Yes (Thermal Discretion) | 6 | 7
  Per Protocol: No (Thermal Discretion) | 0 | 0

9. Secondary Outcome: Protective Sensation Present at 12-months
Description: Summary of Protective Sensation by Month 12
  Semmes-Weinstein Monofilament (SWMF) assessment of protective sensation. The gauge of the monofilaments range from 2.83 (normal) to 6.65 (deep pressure sensation only). Protective Sensation Present (SWMF score of 3.61 or better), Protective Sensation Diminished (SWMF score of 4.31-3.84), Protective Sensation Absent (SWMF score of 4.56 or greater).
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 9
Participants
  modified intent to treat: Protective Sensation Present | 5 | 4
  modified intent to treat: Protective Sensation Diminished | 1 | 3
  modified intent to treat: Protective Sensation Absent | 0 | 2
  per protocol: Protective Sensation Present | 5 | 4
  per protocol: Protective Sensation Diminished | 1 | 3
  per protocol: Protective Sensation Absent | 0 | 2

10. Secondary Outcome: Functional Recovery Classification (Medical Research Council Evaluation of Sensory Function) at 12-months
Description: Summary of Functional Recovery Classification (Medical Research Council Evaluation of Sensory Function) at 12-months
  Patients were assessed for functional recovery of sensation on a scale from S0 to S4 with S0 representing absence of sensibility, S1 representing recovery of deep cutaneous pain sensibility, S2 representing the return of some degree of superficial cutaneous pain and tactile sensibility, S3 representing return of superficial cutaneous pain and tactile sensibility, S3+ representing return of sensibility as in S3 and some recovery of 2-point discrimination (a 2-PD score between 7-15mm), and S4 representing complete recovery of normal sensation as assessed by 2-point discrimination (score between 2-6mm).
Time Frame: 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
Number analyzed (Participants) | 6 | 7
Participants
  modified intent to treat: S1 | 0 | 2
  modified intent to treat: S2 | 0 | 0
  modified intent to treat: S3 | 2 | 0
  modified intent to treat: S3+ | 1 | 0
  modified intent to treat: S4 | 3 | 5
  per protocol: S1 | 0 | 2
  per protocol: S2 | 0 | 0
  per protocol: S3 | 2 | 0
  per protocol: S3+ | 1 | 0
  per protocol: S4 | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of randomization through 1 year.
Arm/Group | Avance Nerve Graft | Hollow Tube Conduit
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/9
Other Adverse Events (participants affected / at risk) | 0/14 | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avance Nerve Graft (N=14) | Hollow Tube Conduit (N=9)
Osteomyleitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2 infection in the affected digit possibly related to the synthetic implant
Infection (Infections and infestations) | 1 (1) | 0 (0) — Infection of grade 2 severity which resulted in prolonged hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avance Nerve Graft (N=14) | Hollow Tube Conduit (N=9)
Occasional Pain (Nervous system disorders) | 0 (0) | 1 (1) — Occasional Pain

LIMITATIONS AND CAVEATS:
1. Early termination due to planned changes in the regulatory status of the study product from an HC/T product to a licensed biologic (planned).
2. High loss-to-follow-up rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No